CLINICAL TRIAL: NCT05166590
Title: Sleep Loss, Cardiovascular Physiology, and Social Experiences Study
Brief Title: Sleep and Social Experiences Study 2
Acronym: SASE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-25169; 5R01HL142051-03 (NIH)
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Sleep; Blood Pressure
Keywords: sleep; heart; stress

STUDY DESIGN:
Intervention Model Description: All participants will be randomized to a night of normal sleep (8 hours) or total sleep restriction.
Who Masked: Participant
Masking Description: Participants will be blind to their condition up until right before they begin their night of normal sleep or total restriction. Participants will also be blind to the nature of the social-rejection task until the debriefing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Sleep (No Intervention): Participants will sleep in the laboratory for 8 hours and then undergo the same social-rejection paradigm as the experimental group to serve as a control comparison.
- Total Sleep Restriction (Experimental): Participants will experience a night of total sleep restriction and then undergo a social-rejection task in the morning.
  Interventions: Behavioral: Sleep Restriction

INTERVENTIONS:
Behavioral: Sleep Restriction — Sleep Deprivation
  Arms: Total Sleep Restriction

SUMMARY:
This study aims to to test effects of sleep loss on perceived discrimination and cardiovascular functioning as well as identify moderators of the racial discrimination and objective sleep link in a sample of 80 African Americans.

DETAILED DESCRIPTION:
African Americans (AAs) are disproportionately burdened by clinical and subclinical cardiovascular disease (CVD) when compared to European Americans (EAs), and while experiences of racial discrimination have been associated with CVD morbidity among AAs, including high daytime and nighttime blood pressure, the mechanisms underlying these associations are unclear. Poor sleep, such as short sleep duration and poor sleep continuity, may serve as a novel pathway; however, this possibility has not been rigorously tested. Evidence linking racial discrimination and poor sleep is mounting, however, largely derived from cross-sectional studies. Further, researchers have largely ignored the possibility of reciprocal effects. In a separate study (CHR#:18-24889) the investigators are testing the effects of perceived discrimination on sleep and nocturnal physiology. In this study, however, the investigators aim to test whether the other direction- whether experimental sleep loss affects one's perception and reaction to social interaction tasks with an outgroup member (White participant). To this end, the investigators will randomize 80 healthy AAs to one night of total sleep restriction or normal sleep in the sleep laboratory and then expose them to several standardized social experience tasks. These tasks include a digit span task, social evaluative speech task and cooperative task (i.e., playing Taboo), all of which will occur in the context of subtle negative evaluative feedback from the White confederate. Cardiovascular functioning as well as self-reported affect will be measured throughout the tasks and potential moderators, including socioeconomic status and race-based rejection sensitivity, will be tested. This study will fill fundamental gap in the scientific literature and provide the critical causal and mechanistic evidence necessary to address racial disparities in sleep and cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to old 64 years old
* Self-identified African American/Black
* English speaking, able to provide informed consent
* Self-reported bedtime between 10 PM and 12 AM for 5/7 nights for the past 3-months (stability to be confirmed by actigraphy and sleep diary)
* Self-reported sleep duration of between 6.5 and 8.5 hours for 5/7 nights for the last month (duration to be confirmed by actigraphy and sleep diary)

Exclusion Criteria:

* Aged greater than 64 years (to minimize age-related differences in sleep quantity and architecture).
* Body mass index of 40 or above (to exclude for obesity, which can impair physiologic recording and confound study outcomes).
* Presence of any clinical sleep disorder, including insomnia and obstructive sleep apnea (OSA), as assessed by validated screening measure. OSA will also be assessed objectively during the Sleep Screening period.
* Medical or psychiatric condition, as assessed by self-report and clinical interview, that is likely to affect sleep/wake function or cardiovascular functioning, including doctor diagnosed arrhythmia, hypertension, congestive heart failure, major depression, bipolar disorder, post-traumatic stress disorder.
* Medication use that is likely to affect sleep/wake function or cardiovascular functioning, including antidepressants, anxiolytic or soporific medication, and beta-blockers.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure post-rejection | Baseline to post final rejection (cooperative task) an average of 32 minutes
  Both systolic and diastolic blood pressure is measured via blood pressure arm cuff, taken after a 5-minute resting period and after each social interaction task

SECONDARY OUTCOMES:
Change in pre-ejection period (PEP) in response to rejection task | Baseline to Post-rejection task, anticipated average of 42 minutes
  Heart rate variability is measured via EKG, averaged over a 5-minute baseline period and in the minutes during the rejection task
Change in heart rate variability (HRV) in response to rejection task | Baseline to Post-rejection task, anticipated average of 42 minutes
  Heart rate variability is measured via EKG, averaged over a 5-minute baseline period and in the minutes during the rejection task
Change in affect | Evening baseline to post-rejection task, time period of approximately 13 hours
  Affect will be measured through the Positive and Negative Affect Scale (PANAS) at multiple timepoints in the study. The PANAS score is calculated by finding the sum of the 10 positive items, and then the 10 negative items. Scores can range from 10-50 for both the Positive and Negative Affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Risk-taking | Immediately after final social rejection task, approximately at hour 13 of the overnight in-lab visit
  Risk-taking post-social rejection will be measured through performance on the Columbia Card Task (hot version), a card game in which they can choose to turn over cards for points. Each card could either be a gain or loss card, but this is unknown until the card is turned over. Turning over gain cards result in point increases while turning over loss cards result in point decreases. Performance is scored by the average number of cards research subjects choose to turn over. Higher average scores (more cards turned over) reflect increased risk-taking. The average is generated across 20 trials of the game, with each trial containing 32 cards in total.
Trust (of outgroup partner) | Public Goods game will be played after the Columbia Card Task, post-social rejection, approximately at hour 13 of the overnight in-lab visit
  Trust (of outgroup partner) will be measured via dollar amount shared in a "common pot" during a Public Goods game. Subjects will be told that they and their outgroup partner have the opportunity to further increase each of their monetary bonus by placing their money in a "common pot" that will be increased by 150% and split equally between them and their partner. Subjects can choose how much they would like to place in the common pot or choose to not share at all. Any money not placed in the common pot will be kept for themselves. Higher amounts (more dollars) shared in the "common pot" indicate higher levels of trust in the outgroup partner.

CONTACTS AND LOCATIONS:
Overall Officials: Aric A Prather, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Our plan is to make all processed data available at the conclusion of the study in line with NIH guidelines.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All processed data should be available within 5 years of completion of the study
Access Criteria: Consistent with NIH guidelines